CLINICAL TRIAL: NCT05341856
Title: Uterine Artery Doppler Changes After Vaginal Administration of Isosorbide Mononitrate In Patients With Unexplained Recurrent Pregnancy Loss
Brief Title: Uterine Artery Doppler Changes After Vaginal Administration of Isosorbide Mononitrate In Patients With URPL
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mostafa Tolba Ahmed, Uterine Artery Doppler Changes After Vaginal Administration of Isosorbide Mononitrate In Patients with Unexplained Recurrent Pregnancy Loss, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: isosorbide mononitrate in URPL
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Recurrent Pregnancy Loss
MeSH Terms: interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uterine artery Doppler Changes After IMN In Patients with URPL (Active Comparator): compare uterine artery blood flow before and after the administration of Isosorbide mononitrate as a nitric oxide donor during mid secretory phase of menstrual cycle for patients with unexplained recurrent pregnancy loss.
  Interventions: Drug: isosorbide mononitrate; Drug: Placebo
- Uterine artery Doppler Changes After placebo In Patients with URPL (Placebo Comparator): compare uterine artery blood flow before and after the administration of placebo during mid secretory phase of menstrual cycle for patients with unexplained recurrent pregnancy loss.
  Interventions: Drug: isosorbide mononitrate; Drug: Placebo

INTERVENTIONS:
Drug: isosorbide mononitrate — insert vaginal tablet of isosorbide mononitrate in cases of unexplained recurrent pregnancy loss
Drug: Placebo — insert vaginal tablet of placebo in cases of unexplained recurrent pregnancy loss

SUMMARY:
compare uterine artery blood flow before and after the administration of Isosorbide mononitrate as a nitric oxide donor during mid secretory phase of menstrual cycle for patients with unexplained recurrent pregnancy loss.

DETAILED DESCRIPTION:
Recurrent pregnancy loss (RPL) is an important reproductive health issue, because it affects 2%-5% of couples. The incidence of RPL varies widely because of the differences in the definitions and criteria used, as well as the populations characteristics (El Hachem et al., 2017).

The reported incidence of early pregnancy loss depends on the method used to detect pregnancy. An estimated 50% of all conceptions are lost at preclinical stages owing to biochemical loss or implantation failure, further 9-20% of clinically recognized pregnancies are miscarried, mainly during the first trimester (weeks 5-12 of gestation), studies consistently demonstrate a sharp reduction after 12 weeks of gestation to an incidence of ~1% suggesting that most pregnancy losses occur soon after implantation (Dimitriadis et al., 2020).

The Royal College of Obstetricians and Gynecologists defines RPL as three or more consecutive pregnancy losses, The most recent RPL guideline from European Society of Human Reproduction and Embryology states that RPL could be considered after the loss of two or more pregnancies and stresses the importance of the need for further scientific research, including epidemiological studies on the effect of various RPL definitions on diagnosis, prognosis and treatment (ESHRE 2017).

Common established causes include uterine anomalies, antiphospholipid syndrome, hormonal and metabolic disorders, and cytogenetic abnormalities. Other etiologies have been proposed but are still considered controversial, such as chronic endometritis, inherited thrombophilia, luteal phase deficiency, and high sperm DNA fragmentation levels (Yang et al., 2019).

Over the years, evidence-based treatments such as surgical correction of uterine anomalies or aspirin and heparin for antiphospholipid syndrome have improved the outcomes for couples with recurrent pregnancy loss. However, almost half of the cases remain unexplained and are empirically treated using progesterone supplementation, anticoagulation, and/or immunomodulatory treatments. Regardless of the cause, the long-term prognosis of couples with recurrent pregnancy loss is good, and most eventually achieve a healthy live birth. However, multiple pregnancy losses can have a significant psychological toll on affected couples, and many efforts are being made to improve treatments and decrease the time needed to achieve a successful pregnancy (El Hachem et al., 2017).

Appropriate endometrial receptivity is vital in achieving a normal pregnancy, Inadequate uterine perfusion leading to endometrial and subendometrial hypoxia could induce low endometrial receptivity, which would increase spontaneous abortion (taylor et al; 2019 & Mansour et al;2020).

Other studies also suggest that uterine perfusion may regulate endometrial receptivity, and that impaired uterine perfusion is one of the causes of URPL. In recent years, Doppler ultrasound with assessments of parameters of uterine artery and endometrium have become widely accepted when evaluating endometrial receptivity(Yang et al., 2019).

Nitric oxide (NO) is a gas and a free radical which is now recognized to have very important physiological roles. NO is important in the endothelium-dependent regulation of blood flow and pressure as well as inhibiting the activation of blood platelets. By this process , NO activates a haem-containing enzyme called soluble guanylyl cyclase which is activated a thousand fold to produce the signaling molecule cyclic GMP. This has many effects at the molecular level to set in train the pathways which propagate the diverse physiological actions of NO(Zhao et al., 2015).

NO plays important functional roles within vascular system, it induce vasodilation ,inhibit platelet aggregation and adhesion to endothelial cells, also inhibit smooth muscle proliferation ,regulates apoptosis and maintain endothelial barrier integrity. NO is the main vasodilator agent in the placenta ,which is the interface between mother and fetus ,and this is the reason why this molecule is crucial in different physiological aspect of pregnancy ,it is involved in implantation ,platelet adhesion ,early embryonic development .Related to placental perfusion, NO seem to influence cytotrophoblastic invasion during first stage of pregnancy and to mediate the remodeling of spiral arteries ,facilitating adequate blood supply to the growing fetus (Zullino et al., 2018).

ELIGIBILITY:
Inclusion Criteria:

* Women age: 20-35 years.

History of recurrent abortion (two or more successive spontaneous abortions) with :

* Normal HSG or hysteroscopy
* Normal serum PRL,
* Normal thyroid function,
* Normal HbA1c,
* Normal pelvic ultrasound
* Negative tests for antiphospholipid antibody syndrome (ACL, Lupus anticoagulant and anti B2 glycoprotein 1) Non pregnant state. Regular menstrual cycles for the previous three months before the study. No hormonal contraception or intrauterine devices. Not on any vasodilator drugs.

Exclusion Criteria:

Age less or more than 20-35. Nulligravidae or nullipara. Infertile women. Induced abortion. Systemic diseases that might affect the hemodynamic indices as thrombocytopenia and thyrotoxicosis.

Cases with uterine anomalies, uterine myomas, polypi and adnexal masses. History of oophorectomy. History of consanguinity. Family history of chromosomal abnormality as Down syndrome and Turner syndrome.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Uterine Artery Doppler Changes After Vaginal Administration of Isosorbide Mononitrate In Patients with Unexplained Recurrent Pregnancy Loss | baseline
  compare uterine artery blood flow before and after the administration of Isosorbide mononitrate as a nitric oxide donor during mid secretory phase of menstrual cycle for patients with unexplained recurrent pregnancy loss.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ali nasr, Professor, Study Director — Al-Azhar University

REFERENCES:
- [Background] Dimitriadis E, Menkhorst E, Saito S, Kutteh WH, Brosens JJ. Recurrent pregnancy loss. Nat Rev Dis Primers. 2020 Dec 10;6(1):98. doi: 10.1038/s41572-020-00228-z. PMID 33303732
- [Background] El Hachem H, Crepaux V, May-Panloup P, Descamps P, Legendre G, Bouet PE. Recurrent pregnancy loss: current perspectives. Int J Womens Health. 2017 May 17;9:331-345. doi: 10.2147/IJWH.S100817. eCollection 2017. PMID 28553146
- [Background] Mansour GM, Hussein SH, Abd El Hady RM, Mohammed HF, Abd El Gawad MM, Abou Gabal AI, Al-Awadhy RM, El Saied M. Uterine artery flow velocity waveform (FVW) type and subednometrial vascularity in recurrent pregnancy loss. J Matern Fetal Neonatal Med. 2020 Feb;33(4):527-532. doi: 10.1080/14767058.2018.1495190. Epub 2018 Aug 6. PMID 29954242
- [Background] Taylor TJ, Quinton AE, de Vries BS, Hyett JA. First-trimester ultrasound features associated with subsequent miscarriage: A prospective study. Aust N Z J Obstet Gynaecol. 2019 Oct;59(5):641-648. doi: 10.1111/ajo.12944. Epub 2019 Feb 6. PMID 30724337
- [Background] Yang W, Wu Z, Yu M, Peng X, Lu W, Feng W, Kang X. Characteristics of midluteal phase uterine artery hemodynamics in patients with recurrent pregnancy loss. J Obstet Gynaecol Res. 2019 Jul;45(7):1230-1235. doi: 10.1111/jog.13944. Epub 2019 Apr 11. PMID 30977230
- [Background] Zhao Y, Vanhoutte PM, Leung SW. Vascular nitric oxide: Beyond eNOS. J Pharmacol Sci. 2015 Oct;129(2):83-94. doi: 10.1016/j.jphs.2015.09.002. Epub 2015 Sep 28. PMID 26499181
- [Background] Zullino S, Buzzella F, Simoncini T. Nitric oxide and the biology of pregnancy. Vascul Pharmacol. 2018 Nov;110:71-74. doi: 10.1016/j.vph.2018.07.004. Epub 2018 Aug 1. PMID 30076925